CLINICAL TRIAL: NCT02611570
Title: Low Dose Computed Tomography Screening Study in Non-smokers with Risk Factors for Lung Cancer in Taiwan
Brief Title: LDCT Screening in Non-smokers in Taiwan
Status: Active, not recruiting | Type: Observational
Sponsor: Academia Sinica, Taiwan (Other)
Collaborators: Taiwan Lung Cancer Society (Other); National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Tri-Service General Hospital (Other); Chang Gung Memorial Hospital (Other); Taichung Veterans General Hospital (Other); Chung Shan Medical University (Other); Kaohsiung Veterans General Hospital. (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); China Medical University Hospital (Other); National Health Research Institutes, Taiwan (Other); Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Principal Investigator, Pan-Chyr Yang, MD, PhD, Research Fellow, Academia Sinica, Taiwan
Other Study IDs: AS-IRB-BM-15039
Record Dates: First submitted 2015-10-26; First posted 2015-11-23 (Estimated); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Low dose computed tomography; Screening; Non-smoker; Gender issue
MeSH Terms: conditions — Lung Neoplasms; Sexism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples Urine samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Non-smokers at risk for lung cancer: 1. Non-smoking subjects with lung cancer family history
  2. Non-smoking subjects with a given lung cancer risk other than lung cancer family history
  Interventions: Other: LDCT

INTERVENTIONS:
Other: LDCT — LDCT at enrollment, annually for two years and biennially for 6 years if no lung cancer is detected

SUMMARY:
This study utilizes the low dose computed tomography(LDCT) to detect the occurrence of early lung cancer among non-smokers in Taiwan. Subjects who have family history of lung cancer or have high risk exposures to lung cancer will be recruited to participate LDCT screening and followed up for their possible occurrence of lung cancer.

DETAILED DESCRIPTION:
Lung cancer ranks the No. 1 lethal cancer in Taiwan, with a five-year survival rate (5-yr SR) of only 15%. Most of the patients with early lung cancer are asymptomatic, while 75% of patients with cancer-related symptom at diagnosis have local or distant metastasis. Compared to a 5-yr SR of 70-90% in stage I/II lung cancer, the 5-yr SR in late stage IIIb/IV is less than 15%. Despite the progress in pharmaceutical treatment for late stage disease, early detection is still the only way to improve the outcome and even cure of this potentially lethal disease. Low dose computed tomography (LDCT) in recognized as the best tool available for early diagnosis of lung cancer. However, the radiation exposure, high cost and high false-positive rate are the major concerns to adapt this detection tool to general population. Recent studies from Europe and US have shown that LDCT screening in high-risk cigarette smoking population can effectively reduce lung cancer mortality. However, the major type of lung cancer in Taiwan is adenocarcinoma, which commonly occurs in non-smoker. Therefore, the risk prediction model generated from studies of western countries may not be suitable for directly adapted to our country. LDCT screening for lung cancer detection in non-smoker remains a controversial issue worldwide, including Taiwan. Facing the unmet need, it is urgent to establish the risk assessment model to predict lung cancer risks in non-smokers and to evaluate the efficacy of LDCT screening in non-smoker high-risk population. In this study, we plan to enroll 12000 non-smoker subjects with a given lung cancer risk; half of them should have lung cancer family history. Each participant will receive LDCT at baseline, annually for two years, and biennially for 6 years. Our overall goal is to establish a risk assessment model of lung cancer in non-smokers and provide suggestions to government for considerations for lung cancer prevention and screening policy in Taiwan.

There are three specific aims in our proposed study:

Aim 1: To evaluate the risk assessment model for predicting lung cancer in non-smokers According to the results of LDCT screening, we expect to improve the risk prediction model for nonsmoker female established by GELAC study. The revised risk model will help recognizing higher risk population.

Aim 2: To establish the protocol for LDCT screening pilot study in Taiwan Establishing working protocol and procedures of LDCT screening to assure a homogeneous behavior among study sites

Aim 3: To establish the efficacy of LDCT screening for lung cancer in non-smoker Lung cancer detection rate, false-positive rate, and cost-effectiveness analysis of LDCT screening for non-smoker lung cancer in Taiwan will be established.

ELIGIBILITY:
Inclusion Criteria:

1. Never smokers or have smoked less than 10 pack-years and quitted smoking over 15 years.
2. age from 55 to 75 years for subjects without lung cancer family history; age 50-75 years for subjects with lung cancer family history (age less than 50 but older than the age at diagnosis of the youngest lung cancer proband is also eligible)
3. Having at least one of the following conditions:

(1)with family history of lung cancer within 1st, 2nd or 3rd degree relatives (2)with exposure history of environmental tobacco smoke in workplace or in home (3)history of chronic lung disease (Tuberculosis or COPD) (4)the cooking index equal or over than 110 [cooking index = 2/7 x (days of cooking by pan frying, stir frying, or deep frying in one week) x (cooking years)] (5)cooking without using cooking ventilation

Exclusion Criteria:

1. with history of lung cancer, or with cancers except skin cancer or cervical carcinoma in situ in the past 5 years
2. can not accept invasive diagnostic procedure or surgery
3. have been examined by chest computed tomography in the past 18 months
4. have unexplained hemoptysis in one month
5. weight loss over than 6 kg with unexplained reason among one year
6. pregnant

Max Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: High risk population for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2014-10; Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Validity of LDCT for lung cancer among non-smokers | 3 years
  True positive, false positive, true negative and false negative rates of LDCT on lung cancer screening. Each subject who is recognized as high risk to lung cancer will be recruited between 2014-2016.

SECONDARY OUTCOMES:
Monitoring the occurrence of lung cancer | 5 years
  Subjects who are recruited between 2014-2016 in this study will be followed every 3-12 months according to their nodule(s) discovered by LDCT for 5 years to obtain their potential occurrence of lung cancer
Monitoring the recurrence of lung cancer | 5 years
  Subjects who have been diagnosed as lung cancer in this study will be monitored for their potential recurrence of lung cancer after clinical treatments/surgery by 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pan-Chyr Yang, M.D., Ph.D., Principal Investigator — National Taiwan University
Locations (17):
- Taiwan (17):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - E-Da Cancer Hospital, Kaohsiung City
  - Shuang-Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Wan Fang Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

REFERENCES:
- [Background] Siegel R, Ma J, Zou Z, Jemal A. Cancer statistics, 2014. CA Cancer J Clin. 2014 Jan-Feb;64(1):9-29. doi: 10.3322/caac.21208. Epub 2014 Jan 7. PMID 24399786
- [Background] International Early Lung Cancer Action Program Investigators; Henschke CI, Yankelevitz DF, Libby DM, Pasmantier MW, Smith JP, Miettinen OS. Survival of patients with stage I lung cancer detected on CT screening. N Engl J Med. 2006 Oct 26;355(17):1763-71. doi: 10.1056/NEJMoa060476. PMID 17065637
- [Background] Field JK, Oudkerk M, Pedersen JH, Duffy SW. Prospects for population screening and diagnosis of lung cancer. Lancet. 2013 Aug 24;382(9893):732-41. doi: 10.1016/S0140-6736(13)61614-1. PMID 23972816
- [Background] Melamed MR, Flehinger BJ, Zaman MB, Heelan RT, Perchick WA, Martini N. Screening for early lung cancer. Results of the Memorial Sloan-Kettering study in New York. Chest. 1984 Jul;86(1):44-53. doi: 10.1378/chest.86.1.44. PMID 6734291
- [Background] Oken MM, Hocking WG, Kvale PA, Andriole GL, Buys SS, Church TR, Crawford ED, Fouad MN, Isaacs C, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Ragard LR, Rathmell JM, Riley TL, Wright P, Caparaso N, Hu P, Izmirlian G, Pinsky PF, Prorok PC, Kramer BS, Miller AB, Gohagan JK, Berg CD; PLCO Project Team. Screening by chest radiograph and lung cancer mortality: the Prostate, Lung, Colorectal, and Ovarian (PLCO) randomized trial. JAMA. 2011 Nov 2;306(17):1865-73. doi: 10.1001/jama.2011.1591. Epub 2011 Oct 26. PMID 22031728
- [Background] Sobue T, Moriyama N, Kaneko M, Kusumoto M, Kobayashi T, Tsuchiya R, Kakinuma R, Ohmatsu H, Nagai K, Nishiyama H, Matsui E, Eguchi K. Screening for lung cancer with low-dose helical computed tomography: anti-lung cancer association project. J Clin Oncol. 2002 Feb 15;20(4):911-20. doi: 10.1200/JCO.2002.20.4.911. PMID 11844811
- [Background] Henschke CI. Early lung cancer action project: overall design and findings from baseline screening. Cancer. 2000 Dec 1;89(11 Suppl):2474-82. doi: 10.1002/1097-0142(20001201)89:11+3.3.co;2-u. PMID 11147630
- [Background] Gohagan J, Marcus P, Fagerstrom R, Pinsky P, Kramer B, Prorok P; Writing Committee, Lung Screening Study Research Group. Baseline findings of a randomized feasibility trial of lung cancer screening with spiral CT scan vs chest radiograph: the Lung Screening Study of the National Cancer Institute. Chest. 2004 Jul;126(1):114-21. doi: 10.1378/chest.126.1.114. PMID 15249451
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] Diederich S, Wormanns D. Impact of low-dose CT on lung cancer screening. Lung Cancer. 2004 Aug;45 Suppl 2:S13-9. doi: 10.1016/j.lungcan.2004.07.997. PMID 15552777
- [Background] Wender R, Fontham ET, Barrera E Jr, Colditz GA, Church TR, Ettinger DS, Etzioni R, Flowers CR, Gazelle GS, Kelsey DK, LaMonte SJ, Michaelson JS, Oeffinger KC, Shih YC, Sullivan DC, Travis W, Walter L, Wolf AM, Brawley OW, Smith RA. American Cancer Society lung cancer screening guidelines. CA Cancer J Clin. 2013 Mar-Apr;63(2):107-17. doi: 10.3322/caac.21172. Epub 2013 Jan 11. PMID 23315954
- [Background] Jaklitsch MT, Jacobson FL, Austin JH, Field JK, Jett JR, Keshavjee S, MacMahon H, Mulshine JL, Munden RF, Salgia R, Strauss GM, Swanson SJ, Travis WD, Sugarbaker DJ. The American Association for Thoracic Surgery guidelines for lung cancer screening using low-dose computed tomography scans for lung cancer survivors and other high-risk groups. J Thorac Cardiovasc Surg. 2012 Jul;144(1):33-8. doi: 10.1016/j.jtcvs.2012.05.060. PMID 22710039
- [Background] Bach PB, Mirkin JN, Oliver TK, Azzoli CG, Berry DA, Brawley OW, Byers T, Colditz GA, Gould MK, Jett JR, Sabichi AL, Smith-Bindman R, Wood DE, Qaseem A, Detterbeck FC. Benefits and harms of CT screening for lung cancer: a systematic review. JAMA. 2012 Jun 13;307(22):2418-29. doi: 10.1001/jama.2012.5521. PMID 22610500
- [Background] Moyer VA; U.S. Preventive Services Task Force. Screening for lung cancer: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2014 Mar 4;160(5):330-8. doi: 10.7326/M13-2771. PMID 24378917
- [Background] Croswell JM, Baker SG, Marcus PM, Clapp JD, Kramer BS. Cumulative incidence of false-positive test results in lung cancer screening: a randomized trial. Ann Intern Med. 2010 Apr 20;152(8):505-12, W176-80. doi: 10.7326/0003-4819-152-8-201004200-00007. PMID 20404381
- [Background] National Lung Screening Trial Research Team; Church TR, Black WC, Aberle DR, Berg CD, Clingan KL, Duan F, Fagerstrom RM, Gareen IF, Gierada DS, Jones GC, Mahon I, Marcus PM, Sicks JD, Jain A, Baum S. Results of initial low-dose computed tomographic screening for lung cancer. N Engl J Med. 2013 May 23;368(21):1980-91. doi: 10.1056/NEJMoa1209120. PMID 23697514
- [Background] Gareen IF, Duan F, Greco EM, Snyder BS, Boiselle PM, Park ER, Fryback D, Gatsonis C. Impact of lung cancer screening results on participant health-related quality of life and state anxiety in the National Lung Screening Trial. Cancer. 2014 Nov 1;120(21):3401-9. doi: 10.1002/cncr.28833. Epub 2014 Jul 25. PMID 25065710
- [Background] Subramanian J, Govindan R. Lung cancer in never smokers: a review. J Clin Oncol. 2007 Feb 10;25(5):561-70. doi: 10.1200/JCO.2006.06.8015. PMID 17290066
- [Background] Couraud S, Zalcman G, Milleron B, Morin F, Souquet PJ. Lung cancer in never smokers--a review. Eur J Cancer. 2012 Jun;48(9):1299-311. doi: 10.1016/j.ejca.2012.03.007. Epub 2012 Mar 28. PMID 22464348
- [Background] Lo YL, Hsiao CF, Jou YS, Chang GC, Tsai YH, Su WC, Chen YM, Huang MS, Chen HL, Yang PC, Chen CJ, Hsiung CA. ATM polymorphisms and risk of lung cancer among never smokers. Lung Cancer. 2010 Aug;69(2):148-54. doi: 10.1016/j.lungcan.2009.11.007. Epub 2009 Dec 11. PMID 20004998
- [Background] Lo YL, Hsiao CF, Jou YS, Chang GC, Tsai YH, Su WC, Chen KY, Chen YM, Huang MS, Hsieh WS, Chen CJ, Hsiung CA. Polymorphisms of MLH1 and MSH2 genes and the risk of lung cancer among never smokers. Lung Cancer. 2011 Jun;72(3):280-6. doi: 10.1016/j.lungcan.2010.10.009. Epub 2010 Nov 19. PMID 21093954
- [Background] Jou YS, Lo YL, Hsiao CF, Chang GC, Tsai YH, Su WC, Chen YM, Huang MS, Chen HL, Chen CJ, Yang PC, Hsiung CA. Association of an EGFR intron 1 SNP with never-smoking female lung adenocarcinoma patients. Lung Cancer. 2009 Jun;64(3):251-6. doi: 10.1016/j.lungcan.2008.09.014. Epub 2008 Nov 20. PMID 19026460
- [Background] Lo YL, Jou YS, Hsiao CF, Chang GC, Tsai YH, Su WC, Chen KY, Chen YM, Huang MS, Hu CY, Chen CJ, Hsiung CA. A polymorphism in the APE1 gene promoter is associated with lung cancer risk. Cancer Epidemiol Biomarkers Prev. 2009 Jan;18(1):223-9. doi: 10.1158/1055-9965.EPI-08-0749. PMID 19124501
- [Background] Samet JM, Avila-Tang E, Boffetta P, Hannan LM, Olivo-Marston S, Thun MJ, Rudin CM. Lung cancer in never smokers: clinical epidemiology and environmental risk factors. Clin Cancer Res. 2009 Sep 15;15(18):5626-45. doi: 10.1158/1078-0432.CCR-09-0376. PMID 19755391
- [Background] Liaw YP, Huang YC, Lien GW. Patterns of lung cancer mortality in 23 countries: application of the age-period-cohort model. BMC Public Health. 2005 Mar 5;5:22. doi: 10.1186/1471-2458-5-22. PMID 15748289
- [Background] Lo YL, Hsiao CF, Chang GC, Tsai YH, Huang MS, Su WC, Chen YM, Hsin CW, Chang CH, Yang PC, Chen CJ, Hsiung CA. Risk factors for primary lung cancer among never smokers by gender in a matched case-control study. Cancer Causes Control. 2013 Mar;24(3):567-76. doi: 10.1007/s10552-012-9994-x. Epub 2012 May 22. PMID 22729933
- [Background] Yamamoto H, Toyooka S, Mitsudomi T. Impact of EGFR mutation analysis in non-small cell lung cancer. Lung Cancer. 2009 Mar;63(3):315-21. doi: 10.1016/j.lungcan.2008.06.021. Epub 2008 Aug 29. PMID 18760859
- [Background] Toyooka S, Matsuo K, Shigematsu H, Kosaka T, Tokumo M, Yatabe Y, Ichihara S, Inukai M, Suehisa H, Soh J, Kiura K, Fong KM, Lee H, Wistuba II, Gazdar AF, Mitsudomi T, Date H. The impact of sex and smoking status on the mutational spectrum of epidermal growth factor receptor gene in non small cell lung cancer. Clin Cancer Res. 2007 Oct 1;13(19):5763-8. doi: 10.1158/1078-0432.CCR-07-0216. PMID 17908966
- [Background] Wang TJ, Zhou BS. Meta-analysis of the potential relationship between exposure to environmental tobacco smoke and lung cancer in nonsmoking Chinese women. Lung Cancer. 1997 Mar;16(2-3):145-50. doi: 10.1016/s0169-5002(96)00624-1. PMID 9152946
- [Background] Fontham ET, Correa P, Reynolds P, Wu-Williams A, Buffler PA, Greenberg RS, Chen VW, Alterman T, Boyd P, Austin DF, et al. Environmental tobacco smoke and lung cancer in nonsmoking women. A multicenter study. JAMA. 1994 Jun 8;271(22):1752-9. PMID 8196118
- [Background] Kirkland LR. Environmental tobacco smoke and lung cancer in nonsmoking women. JAMA. 1995 Feb 15;273(7):519-20. doi: 10.1001/jama.1995.03520310011006. No abstract available. PMID 7837375
- [Background] Nyberg F, Pershagen G. Passive smoking and lung cancer. Accumulated evidence on lung cancer and environmental tobacco smoke. BMJ. 1998 Aug 1;317(7154):347-8; author reply 348. No abstract available. PMID 9729086
- [Background] Hackshaw AK, Law MR, Wald NJ. The accumulated evidence on lung cancer and environmental tobacco smoke. BMJ. 1997 Oct 18;315(7114):980-8. doi: 10.1136/bmj.315.7114.980. PMID 9365295
- [Background] Ko YC, Cheng LS, Lee CH, Huang JJ, Huang MS, Kao EL, Wang HZ, Lin HJ. Chinese food cooking and lung cancer in women nonsmokers. Am J Epidemiol. 2000 Jan 15;151(2):140-7. doi: 10.1093/oxfordjournals.aje.a010181. PMID 10645816
- [Background] Yu IT, Chiu YL, Au JS, Wong TW, Tang JL. Dose-response relationship between cooking fumes exposures and lung cancer among Chinese nonsmoking women. Cancer Res. 2006 May 1;66(9):4961-7. doi: 10.1158/0008-5472.CAN-05-2932. PMID 16651454
- [Background] Kleinerman RA, Wang Z, Wang L, Metayer C, Zhang S, Brenner AV, Zhang S, Xia Y, Shang B, Lubin JH. Lung cancer and indoor exposure to coal and biomass in rural China. J Occup Environ Med. 2002 Apr;44(4):338-44. doi: 10.1097/00043764-200204000-00014. PMID 11977420
- [Background] Brenner DR, Hung RJ, Tsao MS, Shepherd FA, Johnston MR, Narod S, Rubenstein W, McLaughlin JR. Lung cancer risk in never-smokers: a population-based case-control study of epidemiologic risk factors. BMC Cancer. 2010 Jun 14;10:285. doi: 10.1186/1471-2407-10-285. PMID 20546590
- [Background] Clement-Duchene C, Vignaud JM, Stoufflet A, Bertrand O, Gislard A, Thiberville L, Grosdidier G, Martinet Y, Benichou J, Hainaut P, Paris C. Characteristics of never smoker lung cancer including environmental and occupational risk factors. Lung Cancer. 2010 Feb;67(2):144-50. doi: 10.1016/j.lungcan.2009.04.005. Epub 2009 May 21. PMID 19464070
- [Background] Guha N, Merletti F, Steenland NK, Altieri A, Cogliano V, Straif K. Lung cancer risk in painters: a meta-analysis. Environ Health Perspect. 2010 Mar;118(3):303-12. doi: 10.1289/ehp.0901402. Epub 2009 Oct 22. PMID 20064777
- [Background] Chen CL, Hsu LI, Chiou HY, Hsueh YM, Chen SY, Wu MM, Chen CJ; Blackfoot Disease Study Group. Ingested arsenic, cigarette smoking, and lung cancer risk: a follow-up study in arseniasis-endemic areas in Taiwan. JAMA. 2004 Dec 22;292(24):2984-90. doi: 10.1001/jama.292.24.2984. PMID 15613666
- [Background] Alavanja MC, Brownson RC, Boice JD Jr, Hock E. Preexisting lung disease and lung cancer among nonsmoking women. Am J Epidemiol. 1992 Sep 15;136(6):623-32. doi: 10.1093/oxfordjournals.aje.a116542. PMID 1442729
- [Background] Ko YC, Lee CH, Chen MJ, Huang CC, Chang WY, Lin HJ, Wang HZ, Chang PY. Risk factors for primary lung cancer among non-smoking women in Taiwan. Int J Epidemiol. 1997 Feb;26(1):24-31. doi: 10.1093/ije/26.1.24. PMID 9126500
- [Background] Hinds MW, Cohen HI, Kolonel LN. Tuberculosis and lung cancer risk in nonsmoking women. Am Rev Respir Dis. 1982 Jun;125(6):776-8. doi: 10.1164/arrd.1982.125.6.776. PMID 7091889
- [Background] Zheng W, Blot WJ, Liao ML, Wang ZX, Levin LI, Zhao JJ, Fraumeni JF Jr, Gao YT. Lung cancer and prior tuberculosis infection in Shanghai. Br J Cancer. 1987 Oct;56(4):501-4. doi: 10.1038/bjc.1987.233. PMID 2825752
- [Background] Simonsen DF, Farkas DK, Sogaard M, Horsburgh CR, Sorensen HT, Thomsen RW. Tuberculosis and risk of cancer: a Danish nationwide cohort study. Int J Tuberc Lung Dis. 2014 Oct;18(10):1211-9. doi: 10.5588/ijtld.14.0161. PMID 25216835
- [Background] Hubbard R, Venn A, Lewis S, Britton J. Lung cancer and cryptogenic fibrosing alveolitis. A population-based cohort study. Am J Respir Crit Care Med. 2000 Jan;161(1):5-8. doi: 10.1164/ajrccm.161.1.9906062. PMID 10619790
- [Background] Harris JM, Johnston ID, Rudd R, Taylor AJ, Cullinan P. Cryptogenic fibrosing alveolitis and lung cancer: the BTS study. Thorax. 2010 Jan;65(1):70-6. doi: 10.1136/thx.2009.121962. Epub 2009 Dec 8. PMID 19996344
- [Background] Liu Y, Steenland K, Rong Y, Hnizdo E, Huang X, Zhang H, Shi T, Sun Y, Wu T, Chen W. Exposure-response analysis and risk assessment for lung cancer in relationship to silica exposure: a 44-year cohort study of 34,018 workers. Am J Epidemiol. 2013 Nov 1;178(9):1424-33. doi: 10.1093/aje/kwt139. Epub 2013 Sep 15. PMID 24043436
- [Background] Koshiol J, Rotunno M, Consonni D, Pesatori AC, De Matteis S, Goldstein AM, Chaturvedi AK, Wacholder S, Landi MT, Lubin JH, Caporaso NE. Chronic obstructive pulmonary disease and altered risk of lung cancer in a population-based case-control study. PLoS One. 2009 Oct 8;4(10):e7380. doi: 10.1371/journal.pone.0007380. PMID 19812684
- [Background] Schwartz AG, Cote ML, Wenzlaff AS, Van Dyke A, Chen W, Ruckdeschel JC, Gadgeel S, Soubani AO. Chronic obstructive lung diseases and risk of non-small cell lung cancer in women. J Thorac Oncol. 2009 Mar;4(3):291-9. doi: 10.1097/JTO.0b013e3181951cd1. PMID 19190518
- [Background] Nitadori J, Inoue M, Iwasaki M, Otani T, Sasazuki S, Nagai K, Tsugane S. Association between lung cancer incidence and family history of lung cancer: data from a large-scale population-based cohort study, the JPHC study. Chest. 2006 Oct;130(4):968-75. doi: 10.1378/chest.130.4.968. PMID 17035426
- [Background] Zhang Y, Shu XO, Gao YT, Ji BT, Yang G, Li HL, Kilfoy B, Rothman N, Zheng W, Chow WH. Family history of cancer and risk of lung cancer among nonsmoking Chinese women. Cancer Epidemiol Biomarkers Prev. 2007 Nov;16(11):2432-5. doi: 10.1158/1055-9965.EPI-07-0398. PMID 18006933
- [Background] Wu PF, Lee CH, Wang MJ, Goggins WB, Chiang TA, Huang MS, Ko YC. Cancer aggregation and complex segregation analysis of families with female non-smoking lung cancer probands in Taiwan. Eur J Cancer. 2004 Jan;40(2):260-6. doi: 10.1016/j.ejca.2003.08.021. PMID 14728941
- [Background] Matakidou A, Eisen T, Houlston RS. Systematic review of the relationship between family history and lung cancer risk. Br J Cancer. 2005 Oct 3;93(7):825-33. doi: 10.1038/sj.bjc.6602769. PMID 16160696
- [Background] Chen KY, Hsiao CF, Chang GC, Tsai YH, Su WC, Perng RP, Huang MS, Hsiung CA, Chen CJ, Yang PC; GEFLAC Study Group. Hormone replacement therapy and lung cancer risk in Chinese. Cancer. 2007 Oct 15;110(8):1768-75. doi: 10.1002/cncr.22987. PMID 17879370
- [Background] Heiss G, Wallace R, Anderson GL, Aragaki A, Beresford SA, Brzyski R, Chlebowski RT, Gass M, LaCroix A, Manson JE, Prentice RL, Rossouw J, Stefanick ML; WHI Investigators. Health risks and benefits 3 years after stopping randomized treatment with estrogen and progestin. JAMA. 2008 Mar 5;299(9):1036-45. doi: 10.1001/jama.299.9.1036. PMID 18319414
- [Background] Chlebowski RT, Schwartz AG, Wakelee H, Anderson GL, Stefanick ML, Manson JE, Rodabough RJ, Chien JW, Wactawski-Wende J, Gass M, Kotchen JM, Johnson KC, O'Sullivan MJ, Ockene JK, Chen C, Hubbell FA; Women's Health Initiative Investigators. Oestrogen plus progestin and lung cancer in postmenopausal women (Women's Health Initiative trial): a post-hoc analysis of a randomised controlled trial. Lancet. 2009 Oct 10;374(9697):1243-51. doi: 10.1016/S0140-6736(09)61526-9. Epub 2009 Sep 18. PMID 19767090
- [Background] Slatore CG, Chien JW, Au DH, Satia JA, White E. Lung cancer and hormone replacement therapy: association in the vitamins and lifestyle study. J Clin Oncol. 2010 Mar 20;28(9):1540-6. doi: 10.1200/JCO.2009.25.9739. Epub 2010 Feb 16. PMID 20159813
- [Background] Yang SY, Yang TY, Li YJ, Chen KC, Liao KM, Hsu KH, Tsai CR, Chen CY, Hsu CP, Hsia JY, Chuang CY, Tsai YH, Chen KY, Huang MS, Su WC, Chen YM, Hsiung CA, Shen CY, Chang GC, Yang PC, Chen CJ. EGFR exon 19 in-frame deletion and polymorphisms of DNA repair genes in never-smoking female lung adenocarcinoma patients. Int J Cancer. 2013 Jan 15;132(2):449-58. doi: 10.1002/ijc.27630. Epub 2012 Jun 28. PMID 22573488
- [Background] Yang SY, Yang TY, Chen KC, Li YJ, Hsu KH, Tsai CR, Chen CY, Hsu CP, Hsia JY, Chuang CY, Tsai YH, Chen KY, Huang MS, Su WC, Chen YM, Hsiung CA, Shen CY, Chang GC, Yang PC, Chen CJ. EGFR L858R mutation and polymorphisms of genes related to estrogen biosynthesis and metabolism in never-smoking female lung adenocarcinoma patients. Clin Cancer Res. 2011 Apr 15;17(8):2149-58. doi: 10.1158/1078-0432.CCR-10-2045. Epub 2011 Feb 7. PMID 21300759
- [Background] Chen KY, Hsiao CF, Chang GC, Tsai YH, Su WC, Chen YM, Huang MS, Hsiung CA, Chen CJ, Yang PC; GELAC Study Group. EGFR polymorphisms, hormone replacement therapy and lung adenocarcinoma risk: analysis from a genome-wide association study in never-smoking women. Carcinogenesis. 2013 Mar;34(3):612-9. doi: 10.1093/carcin/bgs385. Epub 2012 Dec 13. PMID 23239743
- [Background] Hosgood HD 3rd, Wang WC, Hong YC, Wang JC, Chen K, Chang IS, Chen CJ, Lu D, Yin Z, Wu C, Zheng W, Qian B, Park JY, Kim YH, Chatterjee N, Chen Y, Chang GC, Hsiao CF, Yeager M, Tsai YH, Wei H, Kim YT, Wu W, Zhao Z, Chow WH, Zhu X, Lo YL, Sung SW, Chen KY, Yuenger J, Kim JH, Huang L, Chen YH, Gao YT, Kim JH, Huang MS, Jung TH, Caporaso N, Zhao X, Huan Z, Yu D, Kim CH, Su WC, Shu XO, Kim IS, Bassig B, Chen YM, Cha SI, Tan W, Chen H, Yang TY, Sung JS, Wang CL, Li X, Park KH, Yu CJ, Ryu JS, Xiang Y, Hutchinson A, Kim JS, Cai Q, Landi MT, Lee KM, Hung JY, Park JY, Tucker M, Lin CC, Ren Y, Perng RP, Chen CY, Jin L, Chen KC, Li YJ, Chiu YF, Tsai FY, Yang PC, Fraumeni JF Jr, Seow A, Lin D, Zhou B, Chanock S, Hsiung CA, Rothman N, Lan Q. Genetic variant in TP63 on locus 3q28 is associated with risk of lung adenocarcinoma among never-smoking females in Asia. Hum Genet. 2012 Jul;131(7):1197-203. doi: 10.1007/s00439-012-1144-8. Epub 2012 Feb 25. PMID 22367405
- [Background] Hsiung CA, Lan Q, Hong YC, Chen CJ, Hosgood HD, Chang IS, Chatterjee N, Brennan P, Wu C, Zheng W, Chang GC, Wu T, Park JY, Hsiao CF, Kim YH, Shen H, Seow A, Yeager M, Tsai YH, Kim YT, Chow WH, Guo H, Wang WC, Sung SW, Hu Z, Chen KY, Kim JH, Chen Y, Huang L, Lee KM, Lo YL, Gao YT, Kim JH, Liu L, Huang MS, Jung TH, Jin G, Caporaso N, Yu D, Kim CH, Su WC, Shu XO, Xu P, Kim IS, Chen YM, Ma H, Shen M, Cha SI, Tan W, Chang CH, Sung JS, Zhang M, Yang TY, Park KH, Yuenger J, Wang CL, Ryu JS, Xiang Y, Deng Q, Hutchinson A, Kim JS, Cai Q, Landi MT, Yu CJ, Park JY, Tucker M, Hung JY, Lin CC, Perng RP, Boffetta P, Chen CY, Chen KC, Yang SY, Hu CY, Chang CK, Fraumeni JF Jr, Chanock S, Yang PC, Rothman N, Lin D. The 5p15.33 locus is associated with risk of lung adenocarcinoma in never-smoking females in Asia. PLoS Genet. 2010 Aug 5;6(8):e1001051. doi: 10.1371/journal.pgen.1001051. PMID 20700438
- [Background] Wu X, Wang L, Ye Y, Aakre JA, Pu X, Chang GC, Yang PC, Roth JA, Marks RS, Lippman SM, Chang JY, Lu C, Deschamps C, Su WC, Wang WC, Huang MS, Chang DW, Li Y, Pankratz VS, Minna JD, Hong WK, Hildebrandt MA, Hsiung CA, Yang P. Genome-wide association study of genetic predictors of overall survival for non-small cell lung cancer in never smokers. Cancer Res. 2013 Jul 1;73(13):4028-38. doi: 10.1158/0008-5472.CAN-12-4033. Epub 2013 May 23. PMID 23704207
- [Derived] Chang GC, Chiu CH, Yu CJ, Chang YC, Chang YH, Hsu KH, Wu YC, Chen CY, Hsu HH, Wu MT, Yang CT, Chong IW, Lin YC, Hsia TC, Lin MC, Su WC, Lin CB, Lee KY, Wei YF, Lan GY, Chan WP, Wang KL, Wu MH, Tsai HH, Chian CF, Lai RS, Shih JY, Wang CL, Hsu JS, Chen KC, Chen CK, Hsia JY, Peng CK, Tang EK, Hsu CL, Chou TY, Shen WC, Tsai YH, Tsai CM, Chen YM, Lee YC, Chen HY, Yu SL, Chen CJ, Wan YL, Hsiung CA, Yang PC; TALENT Investigators. Low-dose CT screening among never-smokers with or without a family history of lung cancer in Taiwan: a prospective cohort study. Lancet Respir Med. 2024 Feb;12(2):141-152. doi: 10.1016/S2213-2600(23)00338-7. Epub 2023 Nov 29. PMID 38042167